CLINICAL TRIAL: NCT06183515
Title: The Effect of Continuous Positive Airway Pressure (CPAP) Application on Airway Problems in Pediatric Patients With Subglottic Stenosis Who Undergo Balloon Dilatation
Brief Title: Continuous Positive Airway Pressure (CPAP) Pediatric Patients With Subglottic Stenosis Who Undergo Balloon Dilatation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeliha Alicikus, Head of Anesthesiology and Reanimation department,Assoc Prof, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UERH-AR-ZT-01
Record Dates: First submitted 2023-11-30; First posted 2023-12-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Airway Complication of Anesthesia; Congenital Subglottic Stenosis
Keywords: pediatric airway; subglottic stenosis; apne; CPAP
MeSH Terms: conditions — Laryngostenosis

STUDY DESIGN:
Intervention Model Description: The study included a total of 81 pediatric patients who were 0 to 12 years of age, classified as II and III according to the American Society of Anesthesiologists (ASA), and who underwent elective subglottic balloon dilation under general anesthesia due to acquired or congenital subglottic stenosis.Patients were randomized into two groups through computer-generated randomization into two groups: Group non-CPAP (Control, n=41) and Group CPAP (n=40).During the postoperative period, the CPAP group received Fi02:0.6 and 8 to 12 mmHg of nasal CPAP, or CPAP was initiated through the tracheostomy cannula. The non-CPAP group received Fi02:0.6, and oxygen support was provided at a rate of 3 liters per minute (L/min) either via mask for those who were extubated or through a T-piece for those with a tracheostomy cannula.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-CPAP (Control) (Placebo Comparator): The non-CPAP group received Fi02:0.6, and oxygen support was provided at a rate of 3 liters per minute (L/min) either via mask for those who were extubated or through a T-piece for those with a tracheostomy cannula.
  Interventions: Procedure: CPAP group: postoperative CPAP support, non-CPAP group: oxygen 3 liters per minute (L/min) either via mask for those who were extubated or through a T-piece for those with a trash
- CPAP group (Active Comparator): During the postoperative period, the CPAP group received Fi02:0.6 and 8 to 12 mmHg of nasal CPAP, or CPAP was initiated through the tracheostomy cannula.
  Interventions: Procedure: CPAP group: postoperative CPAP support, non-CPAP group: oxygen 3 liters per minute (L/min) either via mask for those who were extubated or through a T-piece for those with a trash

INTERVENTIONS:
Procedure: CPAP group: postoperative CPAP support, non-CPAP group: oxygen 3 liters per minute (L/min) either via mask for those who were extubated or through a T-piece for those with a trash — The effect of CPAP was prevent atelectasis after apnoeic ventilation during the procedure and to reduce post-procedural airway problems.

SUMMARY:
Nasal continuous positive airway pressure (CPAP) acts as a 'pressure' bridge between spontaneous breathing and controlled mechanical ventilation. As a result, there is an increasing trend in the prophylactic use of nasal CPAP in pediatric patients following high-risk airway procedures to reduce postoperative airway complications. Still, there is no study published on the prophylactic use of balloon dilatation in children with tracheal stenosis.The study hypothesizes that implementing postoperative prophylactic CPAP in pediatric cases with subglottic stenosis undergoing balloon dilation may shorten recovery time and minimize airway complications.

DETAILED DESCRIPTION:
Acquired pediatric subglottic stenosis is reported to have a prevalence of 1-2% . This rate reaches 8.3% in different case series. Acquired pediatric subglottic stenosis is commonly attributed to prolonged intubation, whereas the etiology also involves a history of traumatic or difficult airway. Balloon dilation laryngoplasty is an efficient and safe technique for treating primary and secondary acquired laryngotracheal stenosis. It is successfully applied in these children. Airway surgery typically necessitates a deeper level of anesthesia to control airway reflexes and manage the fluctuations in hemodynamic parameters, which are characteristic of this surgery.

Nevertheless, general anesthesia must be applied several times to patients due to the need for multiple balloon dilatations. At the same time, the procedure also necessitates coping with postoperative complications that may arise. Because alveolar collapse, which is related to general anesthesia, impairs gas exchange by creating a shunt effect, potentially increasing perioperative hypoxemic episodes, which in turn increases the risk for postoperative pulmonary complications. A recent retrospective analysis found that 40.6% of children who underwent balloon dilation experienced desaturation. Additionally, tracheotomy was required in 15.6% of cases, with an equal percentage needing tracheal intubation.

Prophylactic CPAP in pediatric cases has been shown to improve oxygenation by reducing the alveolar-arterial oxygen difference after pediatric laparoscopic surgery. However, it has been proven that CPAP applied after pediatric cardiac surgery has favorable effects on peak expiratory flow.

ELIGIBILITY:
Inclusion Criteria:

* ASA 2-3
* acquired or congenital subglottic stenosis

Exclusion Criteria:

* congenital or acquired diseases of the primary lung or choanal atresia
* younger than 38 gestational weeks
* intubated patients
* congenital cardiac defects

Max Age: 144 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Follow-up of recovery time in patients with CPAP compared to those without CPAP | minutes
  recovery unit time and aldrete score

SECONDARY OUTCOMES:
bronchospasm, the number of desaturation events, intubation, tracheostomy, recovery time, and the need for intensive care | hours
  spo2 below %94 is desaturation

CONTACTS AND LOCATIONS:
Overall Officials: zeliha ZT tuncel, Study Director — Umraniye ERH
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tuncel Z, Goksu S, Deligoz O, Saracoglu KT, Albasha A, Abdallah BM, Saracoglu A. The effect of continuous positive airway pressure (CPAP) application on airway problems in pediatric patients with subglottic stenosis who undergo balloon dilatation. Perioper Med (Lond). 2025 Jan 23;14(1):10. doi: 10.1186/s13741-024-00478-5. PMID 39844310